CLINICAL TRIAL: NCT01196845
Title: Inflammation and Oxidative Stress of Adipose Tissue in Obese and Non-obese Patients Having Sleep Apnea Syndrome
Brief Title: Inflammation and Oxidative Stress of Adipose Tissue in Sleep Apnea Syndrome
Acronym: ADISAS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment difficulty
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Centre Hospitalier Universitaire de Saint Etienne (Other); Hospices Civils de Lyon (Other); University Hospital, Geneva (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 09-CHUG-25; 2009-A00826-51 (Registry Identifier: ID RCB)
Record Dates: First submitted 2010-09-06; First posted 2010-09-09 (Estimated); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Decrease of Inflammation of Adipose Tissue; Sleep Apnea Syndrome
Keywords: adipose tissue; obese patients; inflammation; oxidative stress; sleep apnea syndrome
MeSH Terms: conditions — Sleep Apnea Syndromes; Inflammation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- obese + cPAP (Other): Patients with sleep apnea syndrome will be first randomised in 2 arms according to their obesity. They will be secondly randomised in 2 arms receiving either cPAP treatment or Sham cPAP.
  Interventions: Device: cPAP
- obese + Sham cPAP (Other): Patients with sleep apnea syndrome will be first randomised in 2 arms according to their obesity. They will be secondly randomised in 2 arms receiving either cPAP treatment or Sham cPAP.
  Interventions: Device: cPAP
- non-obese + cPAP (Other): Patients with sleep apnea syndrome will be first randomised in 2 arms according to their obesity. They will be secondly randomised in 2 arms receiving either cPAP treatment or Sham cPAP.
  Interventions: Device: cPAP
- non-obese + Sham cPAP (Other): Patients with sleep apnea syndrome will be first randomised in 2 arms according to their obesity. They will be secondly randomised in 2 arms receiving either cPAP treatment or Sham cPAP.
  Interventions: Device: cPAP

INTERVENTIONS:
Device: cPAP — Patients are randomised in 2 arms : cPAP or sham cPAP
  Arms: obese + cPAP
Device: cPAP — Patients are randomised in 2 arms : cPAP or Sham cPAP
  Arms: obese + Sham cPAP
Device: cPAP — Patients are randomised in 2 arms : cPAP or sham cPAP
  Arms: non-obese + cPAP
Device: cPAP — Patients are randomised in 2 arms : cPAP or sham cPAP
  Arms: non-obese + Sham cPAP

SUMMARY:
The main objective of this study is to evaluate the decrease of inflammation of adipose tissue in obese and non-obese patients having a sleep apnea syndrome and treated or not by continuous positive airway pressure (cPAP).

An interim analysis will be performed when 40 patients will be included.

DETAILED DESCRIPTION:
Inflammation of adipose tissue will be evaluated by RT-PCR on mRNA of pro and anti-inflammatory cytokines (IL-1, IL-6, IL-4, IL-10, IL-12, RANTES, TNFa, leptin, adiponectin, CD68).

ELIGIBILITY:
Inclusion Criteria:

* Male between 18 and 70 years old
* Apnea Hypopnea Index > 30/h and > 5% TST with SaO2 < 90%
* patients obese (BMI > 33kg/m2) or non obese (BMI < 27kg/m2)

Exclusion Criteria:

* Female
* coronary ischemic disease, past history of CVA
* chronic pulmonary disease measured by arterial gasometry (PaO2 < 60mmHg and/or PaCO2 > 45mmHg)
* known hepatic disease
* alcohol consumption > 3 units/day
* sleepiness considered to be dangerous by the investigator
* patient having an hazardous work regarding to awareness
* patient being under anticoagulant, antiplatelet drug or having an active stent or bleeding disorder
* patient having an inflammatory syndrome (C-reactive Protein > 10)
* any allergy to local anaesthetics
* chronic muscle pain
* contraindication to MRI

Ages: 18 Years to 69 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-10-16 (Actual); Primary Completion 2017-02-16 (Actual); Study Completion 2017-02-16 (Actual)

PRIMARY OUTCOMES:
Decrease of inflammation in adipose tissue | 2 months
  Obese and non-obese patients having a sleep apnea syndrome will be treated by cPAP or not (placebo arm). Decrease of inflammation in adipose tissue is expected to be observed in patients treated by cPAP.

SECONDARY OUTCOMES:
Decrease of oxidative stress | 2 months
  Measures of oxidative stress will be done in obese and non-obese patients treated either by cPAP or "Placebo cPAP"
measure of insulin sensitivity | 2 months
  Insulin sensitivity will be measured in obese and non-obese patients treated either by cPAP or "placebo cPAP"
Decrease of systemic inflammation | 2 months
  This measure will be done in obese and non-obese patients treated either by cPAP or "placebo cPAP"
Measure of local hypoxemia of adipose tissue | 2 months
  This measure will be done in obese and non-obese patients treated either by cPAP or "placebo cPAP"
Measure of structural and functional changes in skeletal muscle | 2 months
  This measure will be done in obese and non-obese patients treated either by cPAP or "placebo cPAP"
Measure of vascular adhesion factors modifications and protein synthesis signals modifications | 2 months
  This measure will be done in musculus skeletal of obese and non-obese patients treated either by cPAP or "placebo cPAP"
Decrease in endothelial dysfunction | 2 months
  This measure will be done in obese and non-obese patients treated either by cPAP or "placebo cPAP" and correlated to decrease of inflammation and oxidative stress
Decrease in arterial rigidity | 2 months
  This measure will be done in obese and non-obese patients treated either by cPAP or "placebo cPAP" and correlated to decrease of inflammation and oxidative stress

CONTACTS AND LOCATIONS:
Overall Officials: Jean Louis PEPIN, ProfessorPhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital Grenoble, Grenoble, France

REFERENCES:
- [Background] Baguet JP, Hammer L, Levy P, Pierre H, Launois S, Mallion JM, Pepin JL. The severity of oxygen desaturation is predictive of carotid wall thickening and plaque occurrence. Chest. 2005 Nov;128(5):3407-12. doi: 10.1378/chest.128.5.3407. PMID 16304292
- [Background] Shamsuzzaman AS, Gersh BJ, Somers VK. Obstructive sleep apnea: implications for cardiac and vascular disease. JAMA. 2003 Oct 8;290(14):1906-14. doi: 10.1001/jama.290.14.1906. PMID 14532320
- [Background] Hosogai N, Fukuhara A, Oshima K, Miyata Y, Tanaka S, Segawa K, Furukawa S, Tochino Y, Komuro R, Matsuda M, Shimomura I. Adipose tissue hypoxia in obesity and its impact on adipocytokine dysregulation. Diabetes. 2007 Apr;56(4):901-11. doi: 10.2337/db06-0911. PMID 17395738
- [Background] Marin JM, Carrizo SJ, Vicente E, Agusti AG. Long-term cardiovascular outcomes in men with obstructive sleep apnoea-hypopnoea with or without treatment with continuous positive airway pressure: an observational study. Lancet. 2005 Mar 19-25;365(9464):1046-53. doi: 10.1016/S0140-6736(05)71141-7. PMID 15781100
- [Background] Coughlin SR, Mawdsley L, Mugarza JA, Wilding JP, Calverley PM. Cardiovascular and metabolic effects of CPAP in obese males with OSA. Eur Respir J. 2007 Apr;29(4):720-7. doi: 10.1183/09031936.00043306. Epub 2007 Jan 24. PMID 17251237
- [Background] Lavie L. Obstructive sleep apnoea syndrome--an oxidative stress disorder. Sleep Med Rev. 2003 Feb;7(1):35-51. doi: 10.1053/smrv.2002.0261. PMID 12586529
- [Result] Jullian-Desayes I, Tamisier R, Zarski JP, Aron-Wisnewsky J, Launois-Rollinat SH, Trocme C, Levy P, Joyeux-Faure M, Pepin JL. Impact of effective versus sham continuous positive airway pressure on liver injury in obstructive sleep apnoea: Data from randomized trials. Respirology. 2016 Feb;21(2):378-85. doi: 10.1111/resp.12672. Epub 2015 Nov 16. PMID 26567858